CLINICAL TRIAL: NCT04497805
Title: A Phase 2 Clinical Study to Evaluate The Efficacy and Safety of ALLO-ASC-SHEET in the Subjects With Diabetic Wagner Grade II Foot Ulcers
Brief Title: Clinical Study of ALLO-ASC-SHEET in Subjects With Diabetic Wagner Grade II Foot Ulcers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALLO-ASC-SHEET
Record Dates: First submitted 2020-05-15; First posted 2020-08-04 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALLO-ASC-SHEET (Experimental): ALLO-ASC-SHEET Hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells
  Interventions: Biological: ALLO-ASC-SHEET
- Hydrogel SHEET(Vehicle control) (Placebo Comparator): Vehicle Control Hydrogel sheet without allogenic adipose-derived mesenchymal stem cells
  Interventions: Biological: ALLO-ASC-SHEET

INTERVENTIONS:
Biological: ALLO-ASC-SHEET — Hydrogel sheet containing Allogenic Mesenchymal Stem Cells
  Other Names: Hydrogel sheet containing Allogenic Mesenchymal Stem Cells

SUMMARY:
This is a phase 2 double-blind clinical study to evaluate the efficacy and Safety of ALLO-ASC-SHEET in subjects with Diabetic Wagner Grade II Foot Ulcers, compared to placebo therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 80 years of age.
2. Diagnosed with Type I or Type II diabetes and has Wagner Grade II diabetic foot ulcers for longer than 4 weeks at the time of screening.
3. Foot ulcer located in the plantar or dorsal, with ulcer size between1.5 cm2 and 15 cm2.
4. Ulcer, Graded II by Wagner grade, and extended to muscle periosteum, muscle, tendon, or joint capsule, but not to bone.
5. Ulcer is free of necrotic debris,exhibits no signs of clinical infection.
6. Ulcer area blood circulation meets 1 of the following criteria:

   A. Blood vessels around the ulcer detected by Doppler Test to have biphasic or triphasic flow B. Range of Ankle Brachial Index(ABI) is>0.7 to <1.3 C. Transcutaneous oxygen pressure (TcPO2) >30 mmHg.
7. Is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Ulcer is of non-diabetic pathophysiology.
2. The ulcer has increased or decreased in size by ≥30% during 2 weeks screening period.
3. Patient is currently on higher dose antibiotic therapy as defined by increased dose or change in therapy from the initial treatment regimen at screening to treat index wound infection or patient is on suppressive antibiotic therapy for diabetic foot wound infection.
4. The longest dimension of the index wound exceeds 15 cm at the baseline visit.
5. Patient with skin lesion confirmed by biopsy (when Investigator deems suspicious) and then judged by Investigator to be an etiology other than diabetic foot ulcer (i.e.,example skin cancer in situ, pyoderma).
6. Current evidence of active charcot, osteomyelitis, cellulitis, or evidence of other infection including fever or purulentdrainage from wound site.
7. Is Human Immunodeficiency Virus (HIV) positive
8. Havesevere hepatic deficiencies.
9. Have a glycated hemoglobin A1c (HbA1c) level of >10%.
10. Have an allergic or hypersensitive reaction to bovine-derived proteins or fibrin glue.
11. Have severe renal function insufficiency documented with creatinine greater than 3.0 mg/dL.
12. Pregnant or breast-feeding.
13. Is unwilling to use an "effective" method of contraception during the study.
14. Have evidence of current infection including purulent drainage from the wound site.
15. Have a clinically relevant history of alcohol or drugs abuse.
16. Have postprandialblood sugar >350 mg/dL at screening.
17. Is not able to comply with the study requirements.
18. Is considered by the Investigator to have a significant disease which might impact the study.
19. Is considered not suitable for the study by Investigator.
20. Have a history of malignancy within the last 5 years (except basal cell carcinoma in situ).
21. Is currently or were enrolled in another clinical study within 60 days of screening.
22. Have undergone wound treatments with growth factors, dermal substitutes, or other biological therapies within the last 30 days.
23. Is receiving oral or parenteral corticosteroids (In doses greater than 10 mg per day), any immunosuppressive, or cytotoxic agents with unstable dose prior to 4 weeks from screening.
24. Cannot maintain off-loading process.
25. Panel reactive antibody (PRA) levels ≥ 20% at screening.
26. Venereal Disease Research Laboratory test (VDRL) or RPR positive

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Proportions of subjects who achieved complete wound closure. | During 12 weeks
  Proportions of subjects who achieved complete wound closure during the 12 weeks.

SECONDARY OUTCOMES:
Time to initial complete wound closure between the 2 groups. | During 12 weeks
  Measure the time to initial complete wound closure between the 2 groups.
Changes in wound size compared to baseline between the 2 groups. | During 12 weeks
  Wound size is measured by using eKare 3D Wound Measurement system(Mobile Devices).
Proportions of subjects who achieved complete wound closure between the 2 groups by the classification of wound size. | During 12 weeks
  Proportions of subjects who achieved complete wound closure by the classification of wound size, 1.5~7 cm2 and 7.1~15 cm2 between the 2 groups at every visit.
Proportions of subjects who achieved complete wound closure between the 2 groups by the classification of location of diabetic foot ulcer. | During 12 weeks
  Proportions of subjects who achieved complete wound closure by the classification of location of diabetic foot ulcer, plantar and dorsal between the 2 groups at every visit by post-hoc analysis.
Durability of complete wound closure for the additional 24 weeks. | During 36 weeks
  Durability of complete wound closure for the additional 24 weeks from the initial complete wound closure.
  Wound size is measured by using eKare 3D Wound Measurement system(Mobile Devices).

CONTACTS AND LOCATIONS:
Overall Officials: Yun Jung Choi, PM, Study Director — Anterogen Co., Ltd.
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No